CLINICAL TRIAL: NCT01306396
Title: Investigation on the Preventive Effect of Reduced Fructose Consumption on the Development of Non-alcoholic Fatty Liver Disease in Children in a Long Term Study
Brief Title: Effect of Fructose Reduction on Non-alcoholic Fatty Liver Disease (NAFLD) and Metabolic Syndrome in Overweight Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Hohenheim (Other)
Responsible Party: Dr. Ina Bergheim, University of Hohenheim
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03105084 (IB)
Record Dates: First submitted 2011-02-25; First posted 2011-03-01 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Non-alcoholic Fatty Liver Disease
Keywords: NAFLD; metabolic syndrome; children; fructose
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Other): Based on the daily fructose intake assessed at the beginning of the study, children participating in the intervention group are advised to reduce their daily fructose intake about 50%.
  Interventions: Behavioral: dietary intervention mainly focusing on fructose reduction
- Control group (No Intervention): Families participating in the control group are given only one dietary counseling based on the references of the "DGE" at the beginning of the study if they wish.

INTERVENTIONS:
Behavioral: dietary intervention mainly focusing on fructose reduction — Based on the daily fructose intake assessed at the beginning of the study, children participating in the intervention group are advised to reduce their daily fructose intake by 50%. In the first study year, every three months and in the second study year, every six months, nutritional counseling is repeated in small groups in which parents and children are separately trained.
  Arms: Intervention group

SUMMARY:
The aim of the present study is to find out if a dietary intervention mainly focusing on fructose reduction has a preventive effect on the development and progression of NAFLD and the metabolic syndrome in overweight children.

DETAILED DESCRIPTION:
In the intervention study a total of 100 overweight and 50 normal weight children, aged 5-8 years have to be included. At the beginning, two 24-h dietary recalls are performed to assess nutritional intake and fructose consumption. Anthropometric parameters (body weight and height) are measured to calculate BMI and BMI-SDS of the children. Physical activity during leisure time as well as socio-demographic status and "family background" are assessed using different questionnaires. An ultrasound examination of the liver is performed in all participants for detection of signs of fatty liver. From each child included in the study a fasting blood sample is taken to determine the following blood parameters: ALT, AST, γ-GT, uric acid, blood lipids (TG, HDL, LDL, Total cholesterol), blood alcohol, PAI-1 and endotoxin concentration. A part of the blood sample is used for DNA-analysis. In all children systolic (SBP) and diastolic (DBP) blood pressure are also measured. An oral glucose tolerance test (OGTT) is performed after an overnight fast of 12 h (glucose concentration: 1.75 g/kg body weight, maximum 75g). Simultaneously a glucose hydrogen breath test is performed to assess small intestinal bacterial overgrowth (SIBO). After the check-ups at the beginning of the study, children are divided into two study groups: the intervention group and the control group. Based on the daily fructose intake assessed at the beginning of the study, children participating in the intervention group are advised to reduce their daily fructose intake by 50%. In the first study year, every three months and in the second study year, every six months, nutritional counseling is repeated in small groups in which parents and children are separately trained. If families participating in the control group wish, they receive a dietary counseling based on the references of the "DGE" at the beginning of the study. After the first and the second study year the examinations are repeated in all participants (ultrasound examination only after the second study year).

ELIGIBILITY:
Inclusion Criteria:

* BMI > 90 percentile for overweight children
* BMI < 90 percentile for normal weight children
* no signs of fatty liver (maximal fatty liver grade one or slightly elevated ALT, AST, γ-GT concentrations)
* children with metabolic disorders (prehypertension, high triglyceride, cholesterol or fasting glucose levels) are included with agreement of the pediatrics

Exclusion Criteria:

* liver disease (e.g. steatohepatitis)
* diabetes type 1 and 2
* renal insufficiency
* chronic disease of the gastrointestinal tract
* taking drugs affecting lipid or glucose metabolism

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
prevalence of fatty liver disease | 2 years
  Prevalence of fatty liver disease in ultrasound examination after 2 years
changes in blood lipid concentrations | 1, 2 years
  changes in TG, HDL, LDL, total choelsterol concentrations in serum
changes in blood pressure | 1, 2 years
  changes in systolic (SBP) and diastolic (DBP) blood pressure
changes in glucose metabolism | 1, 2 years
  changes in oral glucose tolerance-test

SECONDARY OUTCOMES:
Changes in small intestinal bacterial overgrowth | 1, 2 years
  changes in glucose hydrogen breath test

CONTACTS AND LOCATIONS:
Overall Officials: Ina Bergheim, Ph.D., Principal Investigator — University of Hohenheim, Dept. of Nutritional Medicine (180 a)
Locations (1):
- University of Hohenheim, Dept. of Nutritional Medicine (180 a), Stuttgart, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Engstler AJ, Aumiller T, Degen C, Durr M, Weiss E, Maier IB, Schattenberg JM, Jin CJ, Sellmann C, Bergheim I. Insulin resistance alters hepatic ethanol metabolism: studies in mice and children with non-alcoholic fatty liver disease. Gut. 2016 Sep;65(9):1564-71. doi: 10.1136/gutjnl-2014-308379. Epub 2015 May 25. PMID 26006114
- [Derived] Maier IB, Ozel Y, Wagnerberger S, Bischoff SC, Bergheim I. Dietary pattern and leisure time activity of overweight and normal weight children in Germany: sex-specific differences. Nutr J. 2013 Jan 15;12:14. doi: 10.1186/1475-2891-12-14. PMID 23320866